CLINICAL TRIAL: NCT02662686
Title: Randomized Multi-centric Prospective Study for the Evaluation of "MitoScore" Marker in the Diagnosis of Embryo Viability in Euploids Embryos.
Brief Title: Study for the Evaluation of "MitoScore" Marker in the Diagnosis of Embryo Viability in Euploids Embryos
Acronym: MitoScore
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Antonio Diez, Product Innovation Leader, Igenomix
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1506-IGX-042-AD
Record Dates: First submitted 2016-01-14; First posted 2016-01-25 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Infertility
Keywords: Embryo Implantation; Mitochondrial genes; Mitochondrial DNA; MitoScore; Embryo selection; Embryo viability; Embryo biomarker; Diagnosis of embryo viability in euploids embryos
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Embryo selection for transfer will be based initially on chromosomally normal embryos and secondly on embryo morphology criteria (specific of IVF lab, as standard practice).
  Interventions: Other: Transfer according to morphological criteria
- MitoScore (Experimental): Embryo selection for transfer will be based initially on chromosomal normality and secondly on the MitoScore value, trying to transfer chromosomally normal embryos which contain the lowest number of mitochondrial DNA copies.
  Interventions: Other: Transfer according to the MitoScore results

INTERVENTIONS:
Other: Transfer according to morphological criteria — Embryos will be analyzed by PGS and mitochondrial score on day 3 or day 5/6 biopsy and transferred on day 5/6, according to morphological criteria (control group).
  Arms: Control
Other: Transfer according to the MitoScore results — Embryos will be analyzed by PGS and mitochondrial score on day 3 or day 5/6 biopsy and transferred on day 5/6, according to the MitoScore results (experimental group).
  Arms: MitoScore

SUMMARY:
The number of copies of mitochondrial genes (mtDNA or "MitoScore") is related to the energy supply of the embryo, which can affect its ability to implant in the maternal uterus.

The objective of this study is to analyse the potential of MitoScore before embryo transfer as a marker to identify and select the embryo with greater capacity of implantation. First of all, chromosomally normal embryos will be selected and mtDNA copies will be quantified. Finally, embryos with less copies of mtDNA will be considered for embryo transfer.

DETAILED DESCRIPTION:
The number of mitochondrial DNA copies (mtDNA) of a chromosomally normal embryo is related to a state of energy, which affects the ability of the embryo to implant in the maternal uterus. There is a decrease in the rate of implantation in euploid embryos containing a high number of mtDNA copies. It is known that after a certain number of mtDNA copies implantation is disrupted even in euploid embryos.

The main purpose of this study is to evaluate the possible relationship between the mtDNA content contained in developing embryos and the result of implantation in order to evaluate the potential of such relationship as a diagnostic tool.

The number of mtDNA copies present in chromosomally normal embryos will be quantified. Subsequently, the transfer of euploid embryos after the randomization will be using either routine morphological or MitoScore criteria.

Study population: women undergoing either IVF or egg donation that go through preimplantation genetic screening (PGS) for different indications, either in day 5/6 or day 3.

This is a triple blinded, randomized, prospective, clinical study where patients with embryos analyzed by PGS in blastocyst stage or day 3 and mitochondrial analysis with day 5/6 transfer, with deferred cycle for those analyzed in day 5/6 and fresh embryo transfer for those analyzed in day 3, will be randomized into two groups:

GROUP A: Embryo selection for transfer will be based initially on chromosomal normality and secondly on embryo morphology criteria (specific for IVF lab).

GROUP B: Embryo selection for transfer will be based initially on chromosomal normality and secondly on the MitoScore value, trying to transfer normal embryos containing the lowest number of mitochondrial DNA copies.

ELIGIBILITY:
* Inclusion Criteria:

  * PGS cycles for different indications
  * Maternal age: ≤40 years old (FIV/ICSI patients)
  * Maternal age: <50 years old (OVODON patients)
  * Spermatocyte concentration: > 2 million of spermatocyte/ml
  * Single embryo transfer

    -≥ 8 oocytes MII
  * Number of Antral Follicules (AFC: ≥10 MII)
* Exclusion Criteria:

  * Detection in the moment of inclusion or previous diagnosis of congenital uterine malformations.
  * Patients with embryo sex selection for those countries in which it is allowed.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1718 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 20 days
Pregnancy rate | 12 days

SECONDARY OUTCOMES:
Miscarriage rate | 9 months
Ongoing pregnancy rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Diez, BS PhD, Principal Investigator — Igenomix; Carlos Simon, MD PhD, Study Director — Igenomix
Locations (11):
- Spain (11):
  - IVI Las Palmas, Las Palmas de Gran Canaria, Las Palmas
  - IVI Madrid, Aravaca, Madrid
  - IVI Bilbao, Leioa, Vizcaya
  - IVI Alicante, Alicante
  - IVI Barcelona, Barcelona
  - IVI Malaga, Málaga
  - IVI Murcia, Murcia
  - IVI Vigo, Pontevedra
  - IVI Sevilla, Seville
  - IVI Valencia, Valencia
  - IVI Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No